CLINICAL TRIAL: NCT06931249
Title: Turkish Version of The Pediatric Anesthesia Emergency Delirium (PAED) Scale: Translation and Cross-Cultural Adaptation
Brief Title: Turkish Version of The Pediatric Anesthesia Emergency Delirium
Acronym: PAED
Status: Active, not recruiting | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Faruk Cicekci, Prof Dr, Selcuk University
Other Study IDs: farukcicekci8; Selcuk University (Other: Selcuk University)
Record Dates: First submitted 2025-03-24; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Emergence Delirium, Anesthesia
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- To make a Turkish version of the English version of the PAED scale, to determine it as a culturally: Translation and cross-cultural adaptation of the PAED scale In Phase 1 (translation), the PAED scale will first be translated into Turkish by three anesthesiologists who are fluent in English.
  In Phase 2 (synthesis), the three translated versions will be combined into a single version.
  In Phase 3 (back translation to English), an English expert who is fluent in Turkish will independently perform the back translation.
  In Phase 4 (expert committee review), the final version of the scale will be evaluated by all raters.
  In Phase 5 (pre-test), anesthesiologists will be contacted through the branch association to ask about the importance and acceptability of the scale in clinical settings and to evaluate the accuracy and comprehensibility of the scale.
  In Phase 6 (Integration), it will be evaluated by all authors and integrated into the final version of the scale.
  Interventions: Behavioral: The observational study

INTERVENTIONS:
Behavioral: The observational study — This study is being conducted to create a Turkish version of the English version of the PAED scale, which did not exist before, and to determine its cultural suitability.

SUMMARY:
Emergence delirium (ED) is a mental disorder seen in children during recovery from general anesthesia. The Pediatric Anesthesia Emergence Delirium (PAED) scale is the only valid scale to assess ED in pediatric patients undergoing general anesthesia. The aim of this study is to translate and adapt the PAED scale to Turkish.

A five-stage translation and adaptation process will be performed. The reliability of the Turkish version of the PAED scale was independently assessed by a group of two raters (anesthesiologists or postanesthesia care unit nurses) in pediatric patients after general anesthesia. ED was defined by a cut-off point of ≥ 10 points on the PAED scale

ELIGIBILITY:
Inclusion Criteria:

1. Parents consented to the study,
2. Transferred to PACU after general anesthesia,
3. Between 2-16 years of age,
4. ASA physical status class I-II,
5. Cognitively intact children.

Exclusion Criteria:

1. Children without parental consent,
2. Children under 2 years of age and over 16 years of age,
3. Children with ASA physical status class III and above,
4. Children who underwent surgery under general anesthesia under emergency conditions,
5. Children with cognitive and behavioral disorders,
6. Children who developed major complications after the operation,
7. Children who are expected to require postoperative mechanical ventilation.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: In patients admitted to the Postoperative Anesthesia Recovery Unit (PACU) after general anesthesia for elective pediatric surgery
Sampling Method: Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Turkish version of the pediatric anesthesia emergency delirium (PAED) scale | 6 months
  The PAED scale consists of the following 5 items; 1- degree of eye contact, 2- purposeful actions, 3- awareness of the environment, 4- restlessness and 5- inconsolability. Each item is assigned a score between 0 and 4,

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://pmc.ncbi.nlm.nih.gov/articles/PMC10387856/pdf/turkjmedsci-52-4-997.pdf